CLINICAL TRIAL: NCT07243470
Title: A Multicenter, Open-label Phase I/II Trial Aiming to Assess the Safety and Clinical Activity of Tarlatamab in Combination With Metronomic Temozolomide in Adolescents and Adults' Patients With High Grade Brain Tumors
Brief Title: Combination of Tarlatamab and Temozolomide in Patients With Central Nervous System Tumors
Acronym: TARLATEM
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: Amgen (Industry); National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ET23-040; 2023-510568-11-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-30; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Glioma; CNS Tumor, Adult; CNS Tumor, Childhood
Keywords: temozolomide; tarlatamab; phase 1/2; RP2D; glioma
MeSH Terms: conditions — Glioma; Central Nervous System Neoplasms | interventions — Temozolomide

STUDY DESIGN:
Intervention Model Description: The study consists of 2 parts:
  A Phase I (safety run-in) part to confirm the safety of tarlatamab single agent followed by combination with a fixed dose of metronomic temozolomide (TMZ).
  Patients start at DL1 with a test dose of tarlatamab 1 mg (C1D1), followed by 10 mg on D8 and D15 of cycle 1 without TMZ. From cycle 2 onward, they receive 10 mg of tarlatamab on D1 and D15 of each 4-week cycle in combination with TMZ.
  Adult safety run in cohort will be opened first, then adolescent safety run in cohort will be evaluated only once the adult safety run in is cleared. A one-week delay period between each pediatric enrolment will be required during pediatric safety run in.
  A Phase II part to assess the clinical activity of the proposed strategy in 3 independent and parallel cohorts: IDH-mutant high-grade glioma, other high-grade glioma, and other high-grade CNS tumors. Enrolment in phase II will be possible only after validation of safety run in in adults then in paediatric patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with IDH-mutant glioma (Experimental): Patients must have histologically confirmed diagnosis of central nervous system (CNS) malignant tumor: IDH-mutant high-grade glioma, other high-grade glioma or other high-grade CNS tumors.
  Interventions: Drug: Tarlatamab; Drug: Temozolomide (TMZ)
- Patients with other glioma (Experimental): Patients must have histologically confirmed diagnosis of central nervous system (CNS) malignant tumor: IDH-mutant high-grade glioma, other high-grade glioma or other high-grade CNS tumors.
  Interventions: Drug: Tarlatamab; Drug: Temozolomide (TMZ)
- Patients with other CNS tumors (Experimental): Patients must have histologically confirmed diagnosis of central nervous system (CNS) malignant tumor: IDH-mutant high-grade glioma, other high-grade glioma or other high-grade CNS tumors.
  Interventions: Drug: Tarlatamab; Drug: Temozolomide (TMZ)

INTERVENTIONS:
Drug: Tarlatamab — At the starting dose (DL1): All patients will receive a step dose (1 mg) on C1D1 administered as a 60-minute intravenous (IV) infusion then 10mg at C1D8 and C1D15 of tarlatamab single agent (no temozolomide administered during cycle 1) then tarlatamab at 10mg every D1 & D15 of each 4-week cycle thereafter in combination with temozolomide from C2D1.
  At DL-1: a cycle period will be 6 weeks with tarlatamab administration every 3 weeks after Cycle 1.
Drug: Temozolomide (TMZ) — At DL1 : Metronomic temozolomide will not be administered during the first cycle. It will be administered from the first day of the second cycle, at a dose of 50 mg/m²/day, continuously.
  At DL-1 : Metronomic temozolomide will not be administered during the first cycle. It will be administered from the first day of the second cycle, at a dose of 50 mg/m²/day, continuously.
  Other Names: Temodal

SUMMARY:
This clinical trial is a 2-phase trial designed to evaluate the safety of tarlatamab in combination with a fixed dose of metronomic temozolomide in adolescents and adults with CNS tumors (stratified into two age-based cohorts), and to assess the clinical activity of this therapeutic strategy in three parallel, histology-defined cohorts (IDH-mutant glioma, other gliomas, and other CNS tumors). A pre-screening to detect DLL3 expression by IHC on archival tumor sample must be performed before the therapeutic part. Only patients with DLL3 positive tumor on IHC can be enrolled in the therapeutic part. This pre-screening must be optimally performed during the ongoing treatment line i.e. before documented progression to not delay treatment starts at time of progression. Tumor samples (surgery or biopsy specimen) will be sent to a central lab for IHC testing.

ELIGIBILITY:
Inclusion Criteria:

I1. Patients aged ≥ 12 years old at time of inform consent signature.

I2. Histologically proven diagnosis of central nervous system (CNS) malignant tumor: IDH-mutant high-grade glioma, other high-grade glioma, or other high-grade CNS tumors.

I3. Tumors expressing DLL3 based on IHC staining performed on archival tumor sample i.e. at least 1+ on IHC [patient with no tumor expression of DLL3 are not eligible].

Note- This pre-screening by IHC should be optimally initiated during an ongoing line of treatment i.e. before documented progression. The ICF1 must be signed before to initiate this pre-screening.

I4. Confirmed progressive or refractory disease after at least one line of standard therapy containing radiotherapy and for which no further effective standard therapy exists.

I5. Evaluable or measurable disease as per iRANO criteria.

I6. Performance status (See Appendix 01):

1. Karnofsky PS for pediatric patients ≥16 years of age ≥ 70%;
2. Lansky PS for patients between 12 and 15y: ≥ 70%;
3. PS ECOG for adult patients: 0 or 1.

I7. Life expectancy ≥ 3 months.

I8. Adequate end organ function according to laboratory values defined below :

Hematologic criteria :

* Peripheral absolute neutrophil count (ANC) ≥1.5 G/L (without growth factor support within 7 days)
* Platelet count ≥ 100 G/L (unsupported for > 7 days)
* Hemoglobin ≥ 9.0 g/dL (unsupported for > 7 days)

Renal and hepatic function :

* Creatinine
* Adult patient: Creatinine clearance as per CKD-EPI > 30 mL/min/1.73 m²
* Pediatric patients: Creatinine <1.5 ULN for age or an estimated glomerular filtration rate (GFR) > 60 mL/min/1.73m2 GFR based on the Schwartz equation (Mian and Schwartz 2017) or as per institutional guidelines
* Total bilirubin ≤1.5 x ULN (≤ 3.0 × ULN for patients with Gilbert's syndrome)
* Alanine aminotransferase (ALAT) ≤ 3 x ULN; aspartate aminotransferase (ASAT) ≤ 3 x ULN Coagulation function : Prothrombin time (PT)/international normalized ratio (INR) and partial thromboplastin time (PTT) or activated partial thromboplastin time (APTT) ≤ 1.5 x ULN. Patients on chronic anticoagulation therapy who do not meet the criteria above may be eligible to enrol after discussion with the Sponsor.

I9. Adequate cardiac function defined by Left ventricular ejection fraction (LVEF) ≥50% at baseline.

I10. Adequate pulmonary function as per investigator judgment and no clinically significant pleural effusion. Pleural effusion managed with indwelling pleural catheter (e.g, PleurX) are allowed.

I11. Availability of a representative formalin-fixed paraffin-embedded (FFPE) sample of tumor tissue (resection or biopsy, archival) with an associated pathology report must be available. This tumor sample must meet the following quality/quantity control criteria: ≥30 % of tumor cells.

I12. Patients must have discontinued all previous anti-cancer treatments (approved or investigational) for CNS treatment with respect of wash-out period at time of C1D1 as shown below:

* Cytotoxic and myelosuppressive chemotherapy : ≥21 days (or ≥42 days if prior nitrosourea)
* Metronomic chemotherapy regimen : ≥21 days or ≥5 half-lives of the treatment with the longest half-life (whichever is shorter)
* Targeted agent : ≥21 days or ≥5 half-lives (whichever is shorter)
* Cellular therapy : ≥42 days for any type of cellular therapy (e.g. modified T cells, NK cells, dendritic cells) agent
* Antibody therapy : ≥21 days after the last infusion except for bevacizumab for which a wash out period of 3 months is requested
* Radiotherapy :
* ≥14 days since small port radiation therapy (i.e. local palliative)
* ≥84 days since large-field radiation therapy (i.e. TBI, craniospinal, whole abdominal, total lung, ≥50% or greater pelvic radiation, ≥50% marrow space)
* ≥42 days for other substantial bone marrow radiation
* Surgery : Major surgery ≥ 21 days. Gastrostomy, ventriculo-peritoneal shunt, endoscopic ventriculostomy, tumor biopsy and insertion of central venous access devices are not considered major surgery, but for these procedures, a 48-hour interval must be maintained before C1D1

I13. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior C1D1 and must agree to use highly effective contraceptive measures starting with the Screening Visit through 6 months after the last dose of study drugs and to not breastfeed during this period. Highly effective contraception is defined in Appendix 02.

I14. Sexually active male must agree to use adequate and appropriate contraception while on study drugs and for 6 months after stopping the study drugs.

I15. Ability to understand and sign informed consent and willingness to comply with the study procedures before study entry and written informed consent from parents/legal representative, patient, and age-appropriate assent before any study-specific screening procedures are conducted according to local, regional or national guidelines.

I16. Covered by a medical insurance.

Exclusion Criteria:

E1. Diagnosis of non-CNS tumor.

E2. Diagnosis of diffuse intrinsic pontine glioma.

E3. Current treatment with bevacizumab.

E4. Prior treatment with a DLL3-directed therapy. Note: Prior treatment with TMZ is not an exclusion criteria.

E5. Neurologically unstable or require increasing doses of corticosteroids during the 7 days before C1D1 or local CNS-directed therapy to control their CNS disease. Note: Patients on low doses of corticosteroids (< 0.25mg/kg/d of prednisolone or equivalent) during the 7 days prior to receiving study drugs are eligible.

E6. Evidence of Grade > 1 recent CNS hemorrhage on the baseline MRI scan.

E7. Bulky tumor on imaging defined as:

i. Tumor with any evidence of uncial herniation or severe midline shift ii. Tumor with diameter of > 6 cm in one dimension on contrast-enhanced MRI iii. Tumor that in the opinion of the investigator shows significant mass effect.

E8. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter drug absorption of oral drugs e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, or malabsorption syndrome)

E9. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to C1D1.

E10. Clinically significant, uncontrolled heart disease (including history of any cardiac arrhythmias, e.g., ventricular, supraventricular, nodal arrhythmias, or conduction abnormality within 6 months of C1D1).

E11. Other malignancy unless this malignancy is not expected to interfere with the evaluation of study endpoints (basal or squamous cell carcinoma of the skin, in-situ carcinoma of the cervix, localized prostate cancer), or with no evidence of disease for ≥ 2 years.

E12.History of hypophysitis or pituitary dysfunction.

E13.History of severe allergic or other hypersensitivity reactions to

* chimeric or humanized antibodies or fusion proteins,
* biopharmaceuticals produced in Chinese hamster ovary cells,
* or any component of the tarlatamab formulation.

E14.Known hypersensitivity to any study drug or component of the formulation or to dacarbazine or TMZ.

E15.Acute and ongoing toxicities from previous therapy that have not resolved to Grade ≤1, except for alopecia, neuropathy, ototoxicity and lab values presented in inclusion criteria.

E16.Arterial thrombosis or a history of pulmonary embolism who need anticoagulants.

E17.Evidence of interstitial lung disease or active, non-infectious pneumonitis.

E18.Recurrent pneumonitis (grade 2 or higher) or grade≥3 immune-mediated adverse events or infusion-related reactions including those that lead to permanent discontinuation while on treatment with immuno-oncology agents.

E19. Live vaccines injection within 4 weeks before C1D1. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever and BCG. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however intranasal influenza vaccines (e.g. Flu-Mist®) are live attenuated vaccines, and are not allowed.

E20. Active autoimmune disease or history of autoimmune disease that required systemic treatment within 2 years of the start of study treatment (i.e., with use of disease-modifying agents or immunosuppressive drugs).

E21. Documentation of:

▪ Active hepatitis B (chronic or acute; defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) unless their HBV is stably controlled on nucleoside analogs (eg entecavir or tenofovir) which will be continued for the duration of the study.

Note: Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. HBV DNA test must be performed in these patients prior to C1D1.

* Active hepatitis C. Patients positive for hepatitis C virus (HCV) antibody are eligible only if PCR is negative for HCV RNA, or
* HIV infection

E22. Prior organ or bone marrow transplant

E23. History or current evidence of any condition, co-morbidity, therapy, any active infections, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.

E24. Pregnant or breastfeeding women.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Phase I : Dose limiting toxicities (DLT) assessed as related at least to tarlatamab, occurring during the first 2 cycles of treatment | From Cycle 1 Day 1 to week 8
  Dose limiting toxicities (DLT) defined as the following adverse event (AE) graded according to NCI CTCAE V5.0 or specific grading system for ICANS and CRS, assessed as related at least to tarlatamab, occurring during the first 2 cycles of treatment (i.e. DLT period is 8 weeks for DL1 or 12 weeks if DL-1 is investigated) : - Any Grade 4 non-laboratory toxicity (including CRS).
  * Any Grade 3 non-laboratory toxicity (including CRS) lasting >7 days despite optimal supportive care and with the following exceptions: Grade 3 fatigue, Grade ≥ 3 Diarrhea/Vomiting/Nausea adequately managed with supportive care measures within 14 days.
  * Grade ≥ 3 ICANS.
  * Any Grade 3 or Grade 4 laboratory value if medical intervention is required or the abnormality persists for >1 week.
  * Febrile neutropenia Grade ≥ 3
  * Grade 4 anemia
  * Any Grade 5 toxicity (i.e., toxic death)
  * Any other significant toxicity deemed by the investigator and/or member of the steering meeting to be dose limiting.
Phase II : To assess the clinical activity of the proposed therapeutic strategy in 3 parallel and independent cohorts of CNS tumors (IDH-mutant glioma, other glioma and other CNS tumors). | 12 weeks from the date of first study drug administration (Cycle 1 Day 1)
  Objective response rate at 12 weeks (ORR-12W) according to immunotherapy Response Assessment for Neuro-Oncology (iRANO) criteria

SECONDARY OUTCOMES:
Evaluation of the Duration of Response (DoR) | From the time of first documented response (Complete Response or Partial Response as per iRANO) until the first documented disease progression or death due to underlying cancer, or censored at the date of the last available tumor assessment
Evaluation of the time to objective response (ToR) | From Cycle 1 Day 1 to first documented objective response
  Time to objective Response is defined as time to first documented objective response (Complete Response or Partial Response as per iRANO) following Cycle 1 Day 1
Evaluation of Disease Control Rate (DCR) | From enrollment to the end of treatment at 12 months
  Disease Control Rate (DCR) will be calculated as the percentage of patients who achieve complete response, partial response, or at least six months of stable disease.
Evaluation of Progression-Free Survival (PFS) | From Cycle 1 Day 1 to the date of the first disease progression or death
  Progression-Free Survival will be measured from C1D1 to the date of the first disease progression or death and will be estimated using the Kaplan-Meier method.
Evaluation of Overall Survival (OS) | From Cycle 1 Day 1 to the date of death from any cause
  Overall survival will be estimated using the Kaplan-Meier method.
To collect nature, incidence and severity of Adverse Events graded using Common Terminology Criteria for Adverse Events (CTCAE) V5.0 or specific grading system for ICANS and CRS [safety and tolerability] | From enrollment to the end of treatment at 12 months
  To characterize the safety and tolerability profile of the proposed therapeutic strategy

OTHER OUTCOMES:
To identify biomarkers predictive of tumor response including DLL3 expression during treatment using descriptive statistics and appropriate multivariate models | From enrollment to the end of treatment at 12 months
  Exploratory analyses in tumor will be performed in an effort to understand the association of DLL3 expression with treatment response. Exploratory data will be summarized using descriptive statistics (e.g. N, medians, inter-quartile range, and mean, standard deviation, minimum and maximum for continuous variables and frequency counts and percentages for categorical variables). The relationship between biomarker and efficacy variables will be assessed using appropriate multivariate models.

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - Institut de Cancérologie de l'Ouest, Angers
  - Hôpital Universitaire d'Angers, Angers
  - CHU de Bordeaux, Bordeaux
  - Hôpital Saint-André, Bordeaux
  - Hôpital Neurologique Pierre Wertheimer, Bron
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital de la Timone, Marseille
  - Hôpitaux Universitaires Pitié Salpêtrière - Charles Foix, Paris
  - IUCT - Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Baruchel S, Diezi M, Hargrave D, Stempak D, Gammon J, Moghrabi A, Coppes MJ, Fernandez CV, Bouffet E. Safety and pharmacokinetics of temozolomide using a dose-escalation, metronomic schedule in recurrent paediatric brain tumours. Eur J Cancer. 2006 Sep;42(14):2335-42. doi: 10.1016/j.ejca.2006.03.023. Epub 2006 Aug 8. PMID 16899365
- [Result] Newlands ES, Stevens MF, Wedge SR, Wheelhouse RT, Brock C. Temozolomide: a review of its discovery, chemical properties, pre-clinical development and clinical trials. Cancer Treat Rev. 1997 Jan;23(1):35-61. doi: 10.1016/s0305-7372(97)90019-0. No abstract available. PMID 9189180
- [Result] Farago A.et al. dynamics of DLL3 and ASCL1 expression in SCLC over disease course. J Thorac Oncol. 2018; 13: S970-S971
- [Result] Longton EB. Excision of the trapezium using a palmar approach. J R Coll Surg Edinb. 1972 Nov;17(6):390-1. No abstract available. PMID 4638131
- [Result] Nicholson HS, Kretschmar CS, Krailo M, Bernstein M, Kadota R, Fort D, Friedman H, Harris MB, Tedeschi-Blok N, Mazewski C, Sato J, Reaman GH. Phase 2 study of temozolomide in children and adolescents with recurrent central nervous system tumors: a report from the Children's Oncology Group. Cancer. 2007 Oct 1;110(7):1542-50. doi: 10.1002/cncr.22961. PMID 17705175
- [Result] Murphy EK. Cases from the past; a look back. AORN J. 1987 Feb;45(2):214-7, 220. doi: 10.1016/s0001-2092(07)68334-3. No abstract available. PMID 3548585
- [Result] Geever RF, Murayama T, Case ME, Giles NH. Rearrangement mutations on the 5' side of the qa-2 gene of Neurospora implicate two regions of qa-1F activator-protein interaction. Proc Natl Acad Sci U S A. 1986 Jun;83(11):3944-8. doi: 10.1073/pnas.83.11.3944. PMID 2940595
- [Result] Grill J, Massimino M, Bouffet E, Azizi AA, McCowage G, Canete A, Saran F, Le Deley MC, Varlet P, Morgan PS, Jaspan T, Jones C, Giangaspero F, Smith H, Garcia J, Elze MC, Rousseau RF, Abrey L, Hargrave D, Vassal G. Phase II, Open-Label, Randomized, Multicenter Trial (HERBY) of Bevacizumab in Pediatric Patients With Newly Diagnosed High-Grade Glioma. J Clin Oncol. 2018 Apr 1;36(10):951-958. doi: 10.1200/JCO.2017.76.0611. Epub 2018 Feb 7. PMID 29412784
- [Result] Broniscer A, Chintagumpala M, Fouladi M, Krasin MJ, Kocak M, Bowers DC, Iacono LC, Merchant TE, Stewart CF, Houghton PJ, Kun LE, Ledet D, Gajjar A. Temozolomide after radiotherapy for newly diagnosed high-grade glioma and unfavorable low-grade glioma in children. J Neurooncol. 2006 Feb;76(3):313-9. doi: 10.1007/s11060-005-7409-5. PMID 16200343
- [Result] Jakacki RI, Cohen KJ, Buxton A, Krailo MD, Burger PC, Rosenblum MK, Brat DJ, Hamilton RL, Eckel SP, Zhou T, Lavey RS, Pollack IF. Phase 2 study of concurrent radiotherapy and temozolomide followed by temozolomide and lomustine in the treatment of children with high-grade glioma: a report of the Children's Oncology Group ACNS0423 study. Neuro Oncol. 2016 Oct;18(10):1442-50. doi: 10.1093/neuonc/now038. Epub 2016 Mar 22. PMID 27006176
- [Result] Patel M, McCully C, Godwin K, Balis FM. Plasma and cerebrospinal fluid pharmacokinetics of intravenous temozolomide in non-human primates. J Neurooncol. 2003 Feb;61(3):203-7. doi: 10.1023/a:1022592913323. PMID 12675312
- [Result] Panetta JC, Kirstein MN, Gajjar A, Nair G, Fouladi M, Heideman RL, Wilkinson M, Stewart CF. Population pharmacokinetics of temozolomide and metabolites in infants and children with primary central nervous system tumors. Cancer Chemother Pharmacol. 2003 Dec;52(6):435-41. doi: 10.1007/s00280-003-0670-4. Epub 2003 Sep 16. PMID 13680158
- [Result] Ostermann S, Csajka C, Buclin T, Leyvraz S, Lejeune F, Decosterd LA, Stupp R. Plasma and cerebrospinal fluid population pharmacokinetics of temozolomide in malignant glioma patients. Clin Cancer Res. 2004 Jun 1;10(11):3728-36. doi: 10.1158/1078-0432.CCR-03-0807. PMID 15173079
- [Result] Omuro A, Chan TA, Abrey LE, Khasraw M, Reiner AS, Kaley TJ, Deangelis LM, Lassman AB, Nolan CP, Gavrilovic IT, Hormigo A, Salvant C, Heguy A, Kaufman A, Huse JT, Panageas KS, Hottinger AF, Mellinghoff I. Phase II trial of continuous low-dose temozolomide for patients with recurrent malignant glioma. Neuro Oncol. 2013 Feb;15(2):242-50. doi: 10.1093/neuonc/nos295. Epub 2012 Dec 14. PMID 23243055
- [Result] Kong DS, Lee JI, Kim JH, Kim ST, Kim WS, Suh YL, Dong SM, Nam DH. Phase II trial of low-dose continuous (metronomic) treatment of temozolomide for recurrent glioblastoma. Neuro Oncol. 2010 Mar;12(3):289-96. doi: 10.1093/neuonc/nop030. Epub 2010 Jan 11. PMID 20167817
- [Result] Banissi C, Ghiringhelli F, Chen L, Carpentier AF. Treg depletion with a low-dose metronomic temozolomide regimen in a rat glioma model. Cancer Immunol Immunother. 2009 Oct;58(10):1627-34. doi: 10.1007/s00262-009-0671-1. Epub 2009 Feb 17. PMID 19221744
- [Result] Kim JT, Kim JS, Ko KW, Kong DS, Kang CM, Kim MH, Son MJ, Song HS, Shin HJ, Lee DS, Eoh W, Nam DH. Metronomic treatment of temozolomide inhibits tumor cell growth through reduction of angiogenesis and augmentation of apoptosis in orthotopic models of gliomas. Oncol Rep. 2006 Jul;16(1):33-9. PMID 16786120
- [Result] Banchi M, Fini E, Crucitta S, Bocci G. Metronomic Chemotherapy in Pediatric Oncology: From Preclinical Evidence to Clinical Studies. J Clin Med. 2022 Oct 24;11(21):6254. doi: 10.3390/jcm11216254. PMID 36362482
- [Result] Tisdale MJ. Antitumor imidazotetrazines--XV. Role of guanine O6 alkylation in the mechanism of cytotoxicity of imidazotetrazinones. Biochem Pharmacol. 1987 Feb 15;36(4):457-62. doi: 10.1016/0006-2952(87)90351-0. PMID 3470008
- [Result] Singh K, Hotchkiss KM, Mohan AA, Reedy JL, Sampson JH, Khasraw M. For whom the T cells troll? Bispecific T-cell engagers in glioblastoma. J Immunother Cancer. 2021 Nov;9(11):e003679. doi: 10.1136/jitc-2021-003679. PMID 34795007
- [Result] Lampson LA. Monoclonal antibodies in neuro-oncology: Getting past the blood-brain barrier. MAbs. 2011 Mar-Apr;3(2):153-60. doi: 10.4161/mabs.3.2.14239. Epub 2011 Mar 1. PMID 21150307
- [Result] Bhojnagarwala PS, O'Connell RP, Park D, Liaw K, Ali AR, Bordoloi D, Cassel J, Tursi NJ, Gary E, Weiner DB. In vivo DNA-launched bispecific T cell engager targeting IL-13Ralpha2 controls tumor growth in an animal model of glioblastoma multiforme. Mol Ther Oncolytics. 2022 Jul 6;26:289-301. doi: 10.1016/j.omto.2022.07.003. eCollection 2022 Sep 15. PMID 36090479
- [Result] Coiffier B, Altman A, Pui CH, Younes A, Cairo MS. Guidelines for the management of pediatric and adult tumor lysis syndrome: an evidence-based review. J Clin Oncol. 2008 Jun 1;26(16):2767-78. doi: 10.1200/JCO.2007.15.0177. PMID 18509186
- [Result] Benjamin JE, Stein AS. The role of blinatumomab in patients with relapsed/refractory acute lymphoblastic leukemia. Ther Adv Hematol. 2016 Jun;7(3):142-56. doi: 10.1177/2040620716640422. Epub 2016 Apr 4. PMID 27247755
- [Result] Ahn MJ, Cho BC, Felip E, Korantzis I, Ohashi K, Majem M, Juan-Vidal O, Handzhiev S, Izumi H, Lee JS, Dziadziuszko R, Wolf J, Blackhall F, Reck M, Bustamante Alvarez J, Hummel HD, Dingemans AC, Sands J, Akamatsu H, Owonikoko TK, Ramalingam SS, Borghaei H, Johnson ML, Huang S, Mukherjee S, Minocha M, Jiang T, Martinez P, Anderson ES, Paz-Ares L; DeLLphi-301 Investigators. Tarlatamab for Patients with Previously Treated Small-Cell Lung Cancer. N Engl J Med. 2023 Nov 30;389(22):2063-2075. doi: 10.1056/NEJMoa2307980. Epub 2023 Oct 20. PMID 37861218
- [Result] Paz-Ares L, Champiat S, Lai WV, Izumi H, Govindan R, Boyer M, Hummel HD, Borghaei H, Johnson ML, Steeghs N, Blackhall F, Dowlati A, Reguart N, Yoshida T, He K, Gadgeel SM, Felip E, Zhang Y, Pati A, Minocha M, Mukherjee S, Goldrick A, Nagorsen D, Hashemi Sadraei N, Owonikoko TK. Tarlatamab, a First-in-Class DLL3-Targeted Bispecific T-Cell Engager, in Recurrent Small-Cell Lung Cancer: An Open-Label, Phase I Study. J Clin Oncol. 2023 Jun 1;41(16):2893-2903. doi: 10.1200/JCO.22.02823. Epub 2023 Jan 23. PMID 36689692
- [Result] Hu B, Nandhu MS, Sim H, Agudelo-Garcia PA, Saldivar JC, Dolan CE, Mora ME, Nuovo GJ, Cole SE, Viapiano MS. Fibulin-3 promotes glioma growth and resistance through a novel paracrine regulation of Notch signaling. Cancer Res. 2012 Aug 1;72(15):3873-85. doi: 10.1158/0008-5472.CAN-12-1060. Epub 2012 Jun 4. PMID 22665268
- [Result] Cooper LA, Gutman DA, Long Q, Johnson BA, Cholleti SR, Kurc T, Saltz JH, Brat DJ, Moreno CS. The proneural molecular signature is enriched in oligodendrogliomas and predicts improved survival among diffuse gliomas. PLoS One. 2010 Sep 3;5(9):e12548. doi: 10.1371/journal.pone.0012548. PMID 20838435
- [Result] Jungk C, Mock A, Exner J, Geisenberger C, Warta R, Capper D, Abdollahi A, Friauf S, Lahrmann B, Grabe N, Beckhove P, von Deimling A, Unterberg A, Herold-Mende C. Spatial transcriptome analysis reveals Notch pathway-associated prognostic markers in IDH1 wild-type glioblastoma involving the subventricular zone. BMC Med. 2016 Oct 26;14(1):170. doi: 10.1186/s12916-016-0710-7. PMID 27782828
- [Result] Menyhart O, Fekete JT, Gyorffy B. Gene expression-based biomarkers designating glioblastomas resistant to multiple treatment strategies. Carcinogenesis. 2021 Jun 21;42(6):804-813. doi: 10.1093/carcin/bgab024. PMID 33754151
- [Result] Maimaiti A, Wang X, Hao Y, Jiang L, Shi X, Pei Y, Feng Z, Kasimu M. Integrated Gene Expression and Methylation Analyses Identify DLL3 as a Biomarker for Prognosis of Malignant Glioma. J Mol Neurosci. 2021 Aug;71(8):1622-1635. doi: 10.1007/s12031-021-01817-7. Epub 2021 Mar 13. PMID 33713320
- [Result] Spino M, Kurz SC, Chiriboga L, Serrano J, Zeck B, Sen N, Patel S, Shen G, Vasudevaraja V, Tsirigos A, Suryadevara CM, Frenster JD, Tateishi K, Wakimoto H, Jain R, Riina HA, Nicolaides TP, Sulman EP, Cahill DP, Golfinos JG, Isse K, Saunders LR, Zagzag D, Placantonakis DG, Snuderl M, Chi AS. Cell Surface Notch Ligand DLL3 is a Therapeutic Target in Isocitrate Dehydrogenase-mutant Glioma. Clin Cancer Res. 2019 Feb 15;25(4):1261-1271. doi: 10.1158/1078-0432.CCR-18-2312. Epub 2018 Nov 5. PMID 30397180
- [Result] Phillips HS, Kharbanda S, Chen R, Forrest WF, Soriano RH, Wu TD, Misra A, Nigro JM, Colman H, Soroceanu L, Williams PM, Modrusan Z, Feuerstein BG, Aldape K. Molecular subclasses of high-grade glioma predict prognosis, delineate a pattern of disease progression, and resemble stages in neurogenesis. Cancer Cell. 2006 Mar;9(3):157-73. doi: 10.1016/j.ccr.2006.02.019. PMID 16530701
- [Result] Jones DT, Mulholland SA, Pearson DM, Malley DS, Openshaw SW, Lambert SR, Liu L, Backlund LM, Ichimura K, Collins VP. Adult grade II diffuse astrocytomas are genetically distinct from and more aggressive than their paediatric counterparts. Acta Neuropathol. 2011 Jun;121(6):753-61. doi: 10.1007/s00401-011-0810-6. Epub 2011 Feb 17. PMID 21327941
- [Result] Noor H, Whittaker S, McDonald KL. DLL3 expression and methylation are associated with lower-grade glioma immune microenvironment and prognosis. Genomics. 2022 Mar;114(2):110289. doi: 10.1016/j.ygeno.2022.110289. Epub 2022 Feb 4. PMID 35124175
- [Result] Saunders LR, Bankovich AJ, Anderson WC, Aujay MA, Bheddah S, Black K, Desai R, Escarpe PA, Hampl J, Laysang A, Liu D, Lopez-Molina J, Milton M, Park A, Pysz MA, Shao H, Slingerland B, Torgov M, Williams SA, Foord O, Howard P, Jassem J, Badzio A, Czapiewski P, Harpole DH, Dowlati A, Massion PP, Travis WD, Pietanza MC, Poirier JT, Rudin CM, Stull RA, Dylla SJ. A DLL3-targeted antibody-drug conjugate eradicates high-grade pulmonary neuroendocrine tumor-initiating cells in vivo. Sci Transl Med. 2015 Aug 26;7(302):302ra136. doi: 10.1126/scitranslmed.aac9459. PMID 26311731
- [Result] Geffers I, Serth K, Chapman G, Jaekel R, Schuster-Gossler K, Cordes R, Sparrow DB, Kremmer E, Dunwoodie SL, Klein T, Gossler A. Divergent functions and distinct localization of the Notch ligands DLL1 and DLL3 in vivo. J Cell Biol. 2007 Jul 30;178(3):465-76. doi: 10.1083/jcb.200702009. PMID 17664336
- [Result] Serth K, Schuster-Gossler K, Kremmer E, Hansen B, Marohn-Kohn B, Gossler A. O-fucosylation of DLL3 is required for its function during somitogenesis. PLoS One. 2015 Apr 9;10(4):e0123776. doi: 10.1371/journal.pone.0123776. eCollection 2015. PMID 25856312
- [Result] Chapman G, Sparrow DB, Kremmer E, Dunwoodie SL. Notch inhibition by the ligand DELTA-LIKE 3 defines the mechanism of abnormal vertebral segmentation in spondylocostal dysostosis. Hum Mol Genet. 2011 Mar 1;20(5):905-16. doi: 10.1093/hmg/ddq529. Epub 2010 Dec 7. PMID 21147753
- [Result] Zhou B, Lin W, Long Y, Yang Y, Zhang H, Wu K, Chu Q. Notch signaling pathway: architecture, disease, and therapeutics. Signal Transduct Target Ther. 2022 Mar 24;7(1):95. doi: 10.1038/s41392-022-00934-y. PMID 35332121
- [Result] Takahashi S, Takahashi M, Tanaka S, Takayanagi S, Takami H, Yamazawa E, Nambu S, Miyake M, Satomi K, Ichimura K, Narita Y, Hamamoto R. A New Era of Neuro-Oncology Research Pioneered by Multi-Omics Analysis and Machine Learning. Biomolecules. 2021 Apr 12;11(4):565. doi: 10.3390/biom11040565. PMID 33921457
- [Result] Lopez-Perez CA, Franco-Mojica X, Villanueva-Gaona R, Diaz-Alba A, Rodriguez-Florido MA, Navarro VG. Adult diffuse midline gliomas H3 K27-altered: review of a redefined entity. J Neurooncol. 2022 Jul;158(3):369-378. doi: 10.1007/s11060-022-04024-5. Epub 2022 May 14. PMID 35567713
- [Result] Grimm SA, Chamberlain MC. Anaplastic astrocytoma. CNS Oncol. 2016 Jul;5(3):145-57. doi: 10.2217/cns-2016-0002. Epub 2016 May 27. PMID 27230974
- [Result] McKinnon C, Nandhabalan M, Murray SA, Plaha P. Glioblastoma: clinical presentation, diagnosis, and management. BMJ. 2021 Jul 14;374:n1560. doi: 10.1136/bmj.n1560. No abstract available. PMID 34261630
- [Result] Brandel MG, Alattar AA, Hirshman BR, Dong X, Carroll KT, Ali MA, Carter BS, Chen CC. Survival trends of oligodendroglial tumor patients and associated clinical practice patterns: a SEER-based analysis. J Neurooncol. 2017 May;133(1):173-181. doi: 10.1007/s11060-017-2430-z. Epub 2017 Apr 24. PMID 28439777
- [Result] Ostrom QT, Patil N, Cioffi G, Waite K, Kruchko C, Barnholtz-Sloan JS. CBTRUS Statistical Report: Primary Brain and Other Central Nervous System Tumors Diagnosed in the United States in 2013-2017. Neuro Oncol. 2020 Oct 30;22(12 Suppl 2):iv1-iv96. doi: 10.1093/neuonc/noaa200. PMID 33123732
- [Result] Louis DN, Perry A, Wesseling P, Brat DJ, Cree IA, Figarella-Branger D, Hawkins C, Ng HK, Pfister SM, Reifenberger G, Soffietti R, von Deimling A, Ellison DW. The 2021 WHO Classification of Tumors of the Central Nervous System: a summary. Neuro Oncol. 2021 Aug 2;23(8):1231-1251. doi: 10.1093/neuonc/noab106. PMID 34185076